CLINICAL TRIAL: NCT02680990
Title: Prehabilitation for Patients With Aggressive Gastrointestinal Cancers Undergoing Neoadjuvant Therapy
Brief Title: Resilience and Exercise in Advanced Cancer Treatment
Acronym: REACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Amanda Cooper, MD, Staff Physician, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002745
Record Dates: First submitted 2015-11-25; First posted 2016-02-12 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Pancreatic Adenocarcinoma; Gastric Adenocarcinoma; Adenocarcinoma of the Gastroesophageal Junction
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise Education (Active Comparator): Distribution of exercise education materials
  Interventions: Other: Exercise Education
- Band Together (Experimental): A strength-training and walking program with or without an exercise partner throughout neoadjuvant therapy.
  Interventions: Behavioral: Band Together

INTERVENTIONS:
Behavioral: Band Together — Band Together is a strength training program utilizing resistance bands with progressively increasing resistance, ranging from 3 to 35 pounds. Sessions are to be completed 3 times a week and involve 3 sets of 6 exercises: 1. chair stands, 2. chest press, 3. shoulder press, 4. arm curls, 5. pulls, and 6. calf raises. In addition, Band Together participants will be asked to work up to a walking goal of 10,000 additional steps per week.
  Other Names: strength training and walking program
  Arms: Band Together
Other: Exercise Education — Education will consist of counseling by the healthcare provider with supplemental handouts from the American College of Sports Medicine and the National Institute on Aging/ National Institutes of Health.
  Arms: Exercise Education

SUMMARY:
This is a pilot study to evaluate the feasibility of, adherence to, and early efficacy of Band Together, a strength-training and walking program (intervention arm) vs. education on the benefits of exercise (control arm) in patients with aggressive gastrointestinal (GI) malignancies (gastric, gastroesophageal, and pancreatic cancer) undergoing neoadjuvant therapy.

DETAILED DESCRIPTION:
A growing body of evidence suggests host resilience (lack of frailty, skeletal muscle reserve, etc.) may impact early healing, recovery following neoadjuvant therapy and surgery, and long-term cancer-free survival. It is well-recognized that resilience is enhanced in individuals with proper diet, sleep habits, and exercise. However, it is unknown whether such resilience can be enhanced by training programs initiated at the time of cancer diagnosis. Although exercise interventions may contribute to these improvements, it is unknown how willing and able these patients are to comply with an exercise regimen during the neoadjuvant therapy period. The aim of this study, therefore, is to evaluate compliance with and the efficacy of Band Together, an exercise program combining strength-training and aerobic exercise, in patients with aggressive GI malignancies undergoing neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. New diagnosis of potentially resectable or borderline resectable pancreatic adenocarcinoma, gastric adenocarcinoma, or adenocarcinoma of the gastroesophageal junction.
3. Patients must be evaluated at the Penn State Hershey Medical Center prior to receiving neoadjuvant chemotherapy or chemoradiation.
4. Patients must be deemed appropriate for neoadjuvant therapy by their treating health care providers.
5. The ability to speak and read English.
6. The ability to provide informed consent.

Exclusion Criteria:

1. Angina (stable or unstable)
2. Paraplegia or quadriplegia
3. Joint or muscle conditions that prevent the patient from being able to grip and or lift resistance bands.
4. Patients who have already started neoadjuvant chemotherapy at other institutions.
5. Presence of metastatic disease.
6. Gastric or pancreatic histologies other than adenocarcinoma.
7. Pregnant women.
8. Prisoners
9. Patients screening positive on the Physical Activity Readiness Questionnaire (PAR-Q)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-12; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Feasibility of Large-Scale Trial: Adherence & Contamination | Throughout the course of neoadjuvant therapy (on average 10-12 weeks)
  The mean adherence rates (percentage of prescribed sessions completed) in the intervention group will be determined based on weekly activity diaries. Activity diaries will be completed by the subject throughout their participation in the study and collected upon the end of participation. The mean contamination rates (completed exercise sessions) in the control group will also be determined based on weekly activity diaries.

SECONDARY OUTCOMES:
Feasibility of a Large-Scale Trial: Eligibility & Willingness to Participate | Completion of neoadjuvant therapy (on average 10-12 weeks)
  Potential subjects will be screened using the Physical Activity Readiness Questionnaire; those who may not be ready to begin an exercise program will be ineligible. The proportion of patients who are PAR-Q ineligible will be compared to the proportion of patients who are eligible based on their PAR-Q results. The proportion of patients who are ineligible due to other exclusion criteria will also be compared. All eligible patients who decline to participate in the study will be asked to provide a reason for their decision; the proportion of potential subjects who decline will be compared to the proportion of subjects who do consent and are eligible.
Exercise Partner Benefits | Completion of neoadjuvant therapy (on average 10-12 weeks)
  The mean adherence rates (percentage of prescribed sessions completed) for subjects in the intervention group who have an exercise partner participate in ≥50% of their exercise sessions will be compared to those of subjects who have an exercise partner for <50% of their exercise sessions.
Change in grip strength and upper body strength as a result of intervention | Enrollment in study and completion of neoadjuvant therapy (on average 10-12 weeks)
  Subjects will be tested before starting neoadjuvant therapy using a dynamometer and a hanging scale, and then again after completing neoadjuvant therapy, to determine if their grip strength and/or upper body strength have changed from baseline.
Assessing the interaction between frailty and the Band Together program | Completion of neoadjuvant therapy (on average 10-12 weeks)
  Frail subjects will be identified using Fried's Frailty Criteria and compared to non-frail subjects using the outcome measures described above.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda B Cooper, MD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State College of Medicine, Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cooper AB, Slack R, Fogelman D, Holmes HM, Petzel M, Parker N, Balachandran A, Garg N, Ngo-Huang A, Varadhachary G, Evans DB, Lee JE, Aloia T, Conrad C, Vauthey JN, Fleming JB, Katz MH. Characterization of Anthropometric Changes that Occur During Neoadjuvant Therapy for Potentially Resectable Pancreatic Cancer. Ann Surg Oncol. 2015 Jul;22(7):2416-23. doi: 10.1245/s10434-014-4285-2. Epub 2014 Dec 18. PMID 25519927
- [Background] Dale W, Hemmerich J, Kamm A, Posner MC, Matthews JB, Rothman R, Palakodeti A, Roggin KK. Geriatric assessment improves prediction of surgical outcomes in older adults undergoing pancreaticoduodenectomy: a prospective cohort study. Ann Surg. 2014 May;259(5):960-5. doi: 10.1097/SLA.0000000000000226. PMID 24096757
- [Background] van de Rest O, van der Zwaluw NL, Tieland M, Adam JJ, Hiddink GJ, van Loon LJ, de Groot LC. Effect of resistance-type exercise training with or without protein supplementation on cognitive functioning in frail and pre-frail elderly: secondary analysis of a randomized, double-blind, placebo-controlled trial. Mech Ageing Dev. 2014 Mar-Apr;136-137:85-93. doi: 10.1016/j.mad.2013.12.005. Epub 2013 Dec 27. PMID 24374288
- [Background] Bollwein J, Diekmann R, Kaiser MJ, Bauer JM, Uter W, Sieber CC, Volkert D. Dietary quality is related to frailty in community-dwelling older adults. J Gerontol A Biol Sci Med Sci. 2013 Apr;68(4):483-9. doi: 10.1093/gerona/gls204. Epub 2012 Oct 12. PMID 23064817